CLINICAL TRIAL: NCT00339768
Title: Randomized Multi-Intervention Trial to Inhibit Precancerous Gastric Lesions in Lingu, Shandong Province, China
Brief Title: A Randomized Multi-Intervention Trial to Inhibit Precancerous Gastric Lesions in Lingu, Shandong Province
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 999995029; OH95-C-N029; NCT00134121 (obsolete NCT alias); NCT01338155 (obsolete NCT alias)
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2019-02-19

CONDITIONS: Precancerous Gastric Lesions
Keywords: Helicobacter Pylori; Gastric Cancer Prevention; Precancerous Gastric Lesions
MeSH Terms: interventions — Amoxicillin; Omeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Amox/omepr (Experimental): 2 weeks; placebo controlled
  Interventions: Drug: Amoxicillin/omeprazole
- Garlic (Experimental): Supplement for 7 years; placebo controlled
  Interventions: Drug: Amoxicillin/omeprazole
- Vitamins (Experimental): Supplement for 7 years; placebo controlled
  Interventions: Drug: Amoxicillin/omeprazole

INTERVENTIONS:
Drug: Amoxicillin/omeprazole — To treat Helicobacter pylori infections. 2 week course of amoxicillin 1gm bid, omeprazole 20mg bid. This factorial trial also investigated a supplement of vitamin C, vitamin E and selenium and a garlic supplement.

SUMMARY:
The Division of Cancer Epidemiology and Genetics is conducting a collaborative randomized multi-intervention trial with the Beijing Institute for Cancer Research to evaluate the etiologic role of Helicobacter pylori, garlic, and certain micronutrients in the multi-step process of gastric carcinogenesis. The primary endpoint will not be cancer, but rather the precancerous lesions severe chronic atrophic gastritis, intestinal metaplasia, and dysplasia. The study is designed to detect a stabilizing or mild decrease in the expected age-related progression of precancerous lesions over the course of the trial. Thus the trial can be considered a study of the potential inhibitors of the process of gastric carcinogenesis. The trial will also provide an evaluation of therapy for H. pylori, including an assessment of reinfection rates, a critical need for formulating strategies for infection control in China and other developing countries. Participating in the trial are approximately 3400 adults aged 35-70 who were part of an ongoing survey of precancerous gastric lesions in 13 Linqu villages in Shandong Province. Linqu appears to be an ideal setting for the trial since stomach cancer rates are among the highes in the world, precancerous gastric lesions are prevalent, and the population is stable and well characterized. These individuals will be randomly assigned (taking H. pylori positivity into account) into 8 intervention groups according to a 2(3) factorial design. The interventions are: 1) initial treatment of H. pylori infection with ameprazole and amoxicillin followed by 2) daily supplementation with a combination of alpha-tocopherol, vitamin C, and selenium; and 3) daily supplementation with garlic extracts. No serious side effects have been seen from any of the interventions to date. The study staff will continue to monitor for possible adverse reactions and the population will receive routine medical care follow-up throughout the course of the trial.

As part of the ongoing study in Linqu, all participants received an endoscopic exam in the fall of 1994. Repeat gastroscopic exams with biopsies at 7 standard gastric sites will be conducted during March to May, 1999 and March to May, 2003 to detect early cancers and to evaluate gasatric mucosal status. The subjects will be categorized according to the most advanced lesions detected in all biopsies and assigned a severity score. The three major endpoints for analysis will be: 1) prevalence of dysplasia or cancer 2) prevalence of sever chronic atrophic gastritis, intestinal metaplasia, dysplasia, or cancer; and 3) average severity score.

DETAILED DESCRIPTION:
The Division of Cancer Epidemiology and Genetics is conducting an 8-year collaborative randomized multi-intervention trial with the Beijing Institute for Cancer Research to evaluate the etiologic role of Helicobacter pylori, garlic, and certain micronutrients in the multi-step process of gastric carcinogenesis. The primary endpoint will not be cancer, but rather the precancerous lesions severe chronic atrophic gastritis, intestinal metaplasia, and dysplasia. The study is designed to detect a stabilizing or mild decrease in the expected age-related progression of precancerous lesions over the course of the trial. Thus the trial can be considered a study of the potential inhibitors of the process of gastric carcinogenesis. The trial will also provide an evaluation of therapy for H. pylori, including an assessment of reinfection rates, a critical need for formulating strategies for infection control in China and other developing countries. Participating in the trial are approximately 3400 adults aged 35-70 who were part of an ongoing survey of precancerous gastric lesions in 13 Linqu villages in Shandong Province. Linqu appears to be an ideal setting for the trial since stomach cancer rates are among the highest in the world, precancerous gastric lesions are prevalent, and the population is stable and well characterized. These individuals will be randomly assigned (taking H. pylori positivity into account) into 8 intervention groups according to a 2(3) factorial design. The interventions are: 1) initial treatment of H. pylori infection with omeprazole and amoxicillin followed by 2) daily supplementation with a combination of alpha-tocopherol, vitamin C, and selenium; and 3) daily supplementation with garlic extracts. Compliance was excellent and no serious side effects were seen from any of the interventions.

As part of the ongoing study in Linqu, all participants received an endoscopic exam in the fall of 1994. Repeat gastroscopic exams with biopsies at 7 standard gastric sites conducted during March to May, 1999 and March to April, 2003 to detect early cancers and to evaluate gastric mucosal status. The subjects will be categorized according to the most advanced lesions detected in all biopsies and assigned a severity score. The three major endpoints for analysis will be: 1) prevalence of dysplasia or cancer 2) prevalence of severe chronic atrophic gastritis, intestinal metaplasia, dysplasia, or cancer; and 3) average severity score.

The major endpoint paper was published in JNCI in 2006. Additional analyses of the trial data are underway. A continuation study is proceeding that will allow for follow-up of the approximately 3070 remaining trial participants through 2010 on the long-term effects of the previous treatments on gastric cancer incidence and on cause-specific death rates and allow approximately 364 participants in the previous study with advanced gastric lesions in 2003 an opportunity for annual endoscopic screening for gastric cancer.

ELIGIBILITY:
* INCLUSION CRITERIA:

Ages 35-670 in the 14 Linqu villages who received endoscopy examinations in the fall of 1994.

Both men and women will be included.

Patients must sign an informed consent form indicating a willingness to participate in the 42-month trial.

Must be free of debilitating chronic disease.

Must not report allergies to penicillin or similar medications.

Must not have had previous treatment for H. pylori.

Must not have a history of bleeding disorder.

Must not be taking vitamin/mineral supplements on a regular basis.

EXCLUSION CRITERIA:

Persons with cancer (except resected non-melanotic skin cancer), heart failure, emphysema, and other life-threatening illness will be excluded.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3411 (Actual)
Dates: Start 1995-07-01; Primary Completion 1996-06-10 (Actual); Study Completion 1996-06-10 (Actual)

PRIMARY OUTCOMES:
Precancerous gastric lesions | 7 years
  prevention of cancer
Gastric cancer incidence | 15 years
  prevention of caner

SECONDARY OUTCOMES:
Side effects | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell H Gail, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Beijing Institute for Cancer Research, Beijing, China

REFERENCES:
- [Background] Correa P. Human gastric carcinogenesis: a multistep and multifactorial process--First American Cancer Society Award Lecture on Cancer Epidemiology and Prevention. Cancer Res. 1992 Dec 15;52(24):6735-40. PMID 1458460
- [Background] You WC, Blot WJ, Chang YS, Ershow AG, Yang ZT, An Q, Henderson B, Xu GW, Fraumeni JF Jr, Wang TG. Diet and high risk of stomach cancer in Shandong, China. Cancer Res. 1988 Jun 15;48(12):3518-23. PMID 3370645
- [Background] You WC, Blot WJ, Li JY, Chang YS, Jin ML, Kneller R, Zhang L, Han ZX, Zeng XR, Liu WD, et al. Precancerous gastric lesions in a population at high risk of stomach cancer. Cancer Res. 1993 Mar 15;53(6):1317-21. PMID 8443811
- [Derived] Su XQ, Yin ZY, Jin QY, Liu ZC, Han X, Hu ZQ, Zhang L, Ma JL, Li ZX, Zhang Y, Zhou T, Liu WD, You WC, Pan KF, Shi L, Li WQ. Allium vegetable intake associated with the risk of incident gastric cancer: a continuous follow-up study of a randomized intervention trial. Am J Clin Nutr. 2023 Jan;117(1):22-32. doi: 10.1016/j.ajcnut.2022.10.017. Epub 2022 Dec 20. PMID 36789941
- [Derived] Guo Y, Li ZX, Zhang JY, Ma JL, Zhang L, Zhang Y, Zhou T, Liu WD, Han ZX, Li WQ, Pan KF, You WC. Association Between Lifestyle Factors, Vitamin and Garlic Supplementation, and Gastric Cancer Outcomes: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2020 Jun 1;3(6):e206628. doi: 10.1001/jamanetworkopen.2020.6628. PMID 32589229
- [Derived] Li WQ, Zhang JY, Ma JL, Li ZX, Zhang L, Zhang Y, Guo Y, Zhou T, Li JY, Shen L, Liu WD, Han ZX, Blot WJ, Gail MH, Pan KF, You WC. Effects of Helicobacter pylori treatment and vitamin and garlic supplementation on gastric cancer incidence and mortality: follow-up of a randomized intervention trial. BMJ. 2019 Sep 11;366:l5016. doi: 10.1136/bmj.l5016. PMID 31511230